CLINICAL TRIAL: NCT06568094
Title: An Open, Multicenter Phase Ib/II Study on the Safety, Tolerability and Efficacy of HRS-5041 Tablets Combined With Antitumor Therapy in Subjects With Advanced Prostate Cancer
Brief Title: A Study of HRS-5041 Tablets Combined With Antitumor Therapy in Subjects With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5041-201
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Docetaxel

STUDY DESIGN:
Intervention Model Description: HRS-5041 tablets combined with antitumor therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-5041 tablets combined with Abiraterone Acetate tablets（II）and Prednisone Acetate tablets (Experimental)
  Interventions: Drug: HRS-5041 tablets; Drug: Abiraterone Acetate tablets（II）; Drug: Prednisone Acetate tablets
- HRS-5041 tablets combined with Docetaxel injection and Prednisone Acetate tablets (Experimental)
  Interventions: Drug: HRS-5041 tablets; Drug: Prednisone Acetate tablets; Drug: Docetaxel Injection
- HRS-5041 tablets combined with HRS-1167 tablets (Experimental)
  Interventions: Drug: HRS-5041 tablets; Drug: HRS-1167 tablets
- HRS-5041 tablets combined with SHR2554 tablets (Experimental)
  Interventions: Drug: HRS-5041 tablets; Drug: SHR2554 tablets

INTERVENTIONS:
Drug: HRS-5041 tablets — HRS-5041 tablets
Drug: Abiraterone Acetate tablets（II） — Abiraterone Acetate tablets（II）
  Arms: HRS-5041 tablets combined with Abiraterone Acetate tablets（II）and Prednisone Acetate tablets
Drug: Prednisone Acetate tablets — Prednisone Acetate tablets
  Arms: HRS-5041 tablets combined with Abiraterone Acetate tablets（II）and Prednisone Acetate tablets; HRS-5041 tablets combined with Docetaxel injection and Prednisone Acetate tablets
Drug: Docetaxel Injection — Docetaxel Injection
  Arms: HRS-5041 tablets combined with Docetaxel injection and Prednisone Acetate tablets
Drug: HRS-1167 tablets — HRS-1167 tablets
  Arms: HRS-5041 tablets combined with HRS-1167 tablets
Drug: SHR2554 tablets — SHR2554 tablets
  Arms: HRS-5041 tablets combined with SHR2554 tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy, and safety of HRS-5041 tablets combined with antitumor therapy in subjects with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, and are willing and able to comply with planned visits for medical examinations and other procedural requirements.
2. The age is above 18 years old when signing the informed consent (the ceiling age is 80 years old in the dose escalation phase), male.
3. ECOG score is 0 or 1.
4. An expected survival of ≥ 12 weeks.
5. Adenocarcinoma of the prostate confirmed with histologically or cytologically ,and without a diagnosis of neuroendocrine or small cell carcinoma.
6. Adequate blood samples should be provided for gene mutation detection during the screening period. It is recommended to provide tumor tissue samples.
7. Male subjects whose partner is women of childbearing potential (WOCBP) are required to use highly effective contraception from the date of signing the informed consent until 3 months after the last dose of the investigational drug.

Exclusion Criteria:

1. Plan to receive any other antitumor therapy during this study.
2. Had history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML); Or had other malignancies in the 5 years prior to the first dose.
3. Participants who are participating in another clinical study or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or five half-lives of the investigational drug, whichever is shorter.
4. Had undergone major surgery within 28 days prior to first dosing; Minor traumatic surgery within 7 days prior to first dosing; There are non-healing wounds, untreated fractures.
5. Drugs with a strong inducer or inhibitor of the metabolic enzyme CYP3A have been used in the past, and the washout period from the end time to the first administration in this study is shorter than the 5 half-life of the drug.
6. The toxicity from previous anti-tumor treatment has not recovered to ≤ grade I.
7. Central nervous system or meningeal metastasis of tumors is known or subjects have a history of primary central nervous system tumors.
8. Severe cerebrovascular disease occurred within 6 months prior to administration.
9. Subjects with poorly controlled hypertension and a history of hypertensive crisis or hypertensive encephalopathy.
10. Severe bone injury due to bone metastases, pathological fractures , and spinal cord compression as determined by the investigators at important sites that occurred within the last 6 months or are expected to occur in the near future.
11. Having one of multiple factors that affect the oral drug or having an active gastrointestinal disease or other disease that may significantly affect drug absorption, distribution, metabolism, or excretion.
12. Had history of allergy to the proposed investigational drug or its excipient components.
13. Presence of active heart disease in the 6 months prior to first dosing, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and medically treatable ventricular arrhythmias.
14. Presence of active hepatitis B and hepatitis C; Or serious infected persons requiring antibiotics, antivirals or antifungal drugs to control.
15. Presence of the history of immunodeficiency or organ transplantation.
16. Presence of other serious physical or mental diseases or laboratory abnormalities.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (Phase Ib) | 21 or 28 days
Incidence and severity of adverse events (AE) (Phase Ib) | 2 years
PSA response rate (Phase II) | 1 year

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
Disease control rate (DCR) | 1 year
Duration of response (DoR) | 1 year
PSA response rate | 1 year
Time to PSA progression | 1 year
Radiographic progression-free survival (rPFS) | 1 year
Overall survival (OS) | 2 years
Blood concentrations of HRS-5041(Phase Ib) | 16 weeks
Blood concentrations of HRS-1167(Phase Ib) | 16 weeks
Blood concentrations of SHR2554(Phase Ib) | 16 weeks
Blood concentrations of Abiraterone (Phase Ib) | 16 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Shanghai Jiao Tong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided